CLINICAL TRIAL: NCT01785836
Title: An Extension Study to Assess the Safety, Tolerability, Efficacy, and Treatment Adherence of Dapsone in Acne Vulgaris
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never initiated due to company decision. No study subjects were ever enrolled or dosed.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 225678-005
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapsone Formulation A (Experimental): Dapsone Formulation A applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Interventions: Drug: Dapsone Formulation A
- Dapsone Formulation B (Experimental): Dapsone Formulation B applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Interventions: Drug: Dapsone Formulation B
- Dapsone Formulation C (Experimental): Dapsone Formulation C applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Interventions: Drug: Dapsone Formulation C
- Dapsone 5% Gel (Active Comparator): Dapsone 5% gel (ACZONE®) applied twice daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Interventions: Drug: Dapsone 5% Gel

INTERVENTIONS:
Drug: Dapsone Formulation A — Dapsone Formulation A applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Arms: Dapsone Formulation A
Drug: Dapsone Formulation B — Dapsone Formulation B applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Arms: Dapsone Formulation B
Drug: Dapsone Formulation C — Dapsone Formulation C applied once daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Arms: Dapsone Formulation C
Drug: Dapsone 5% Gel — Dapsone 5% gel (ACZONE®) applied twice daily to the face and upper chest, upper back, and shoulders (as per protocol) for 12 weeks.
  Other Names: ACZONE®
  Arms: Dapsone 5% Gel

SUMMARY:
This study will assess the safety, tolerability, and efficacy of dapsone in subjects with acne vulgaris following 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Allergan study 225678-004

Exclusion Criteria:

* Anticipates the need for surgery or hospitalization during the study

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Inflammatory Lesion Count | Baseline, Week 12

SECONDARY OUTCOMES:
Change from Baseline in Non-Inflammatory Lesion Count | Baseline, Week 12
Change from Baseline in Total Lesion Count | Baseline, Week 12
Percentage of Subjects With a Global Acne Assessment Score (GAAS) of 0 or 1 | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan